CLINICAL TRIAL: NCT04212663
Title: A Multicenter Study on the Treatment of Recurrent Clubfoot With the Tendon Release of Musculi Tibialis Posterior
Brief Title: A Study on the Treatment of Recurrent Clubfoot With the Tendon Release of Musculi Tibialis Posterior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Hongwen Xu, The director of pediatric orthopedic depatment, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuangzhouWCMC-002
Record Dates: First submitted 2019-09-21; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Recurrent Clubfoot
Keywords: Musculi tibialis posterior; Tendon release; Anterior tibial tendon transfer
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): receive the procure of Anterior tibial tendon transfer(TATT) + Achilles tendon lengthing + fascial release
  Interventions: Procedure: Anterior tibial tendon transfer(TATT); Procedure: Achilles tendon lengthing; Procedure: Fascial release
- experiment (Experimental): receive the procure of Anterior tibial tendon transfer(TATT) + Achilles tendon lengthing + fascial release+ The tendon release of musculi tibialis posterior
  Interventions: Procedure: The tendon release of musculi tibialis posterior; Procedure: Anterior tibial tendon transfer(TATT); Procedure: Achilles tendon lengthing; Procedure: Fascial release

INTERVENTIONS:
Procedure: The tendon release of musculi tibialis posterior — To release the tendon of musculi tibialis posterior.
  Arms: experiment
Procedure: Anterior tibial tendon transfer(TATT) — To transfer the the tendon of anterior tibial from the navicular to the third cuneiform.
Procedure: Achilles tendon lengthing — To lengthen the achilles tendon by using two incisions.
Procedure: Fascial release — To cut off the metatarsal fascia in the middle part.

SUMMARY:
The musculi tibialis posterior can adduct the foot, so releasing the tedon of the muscle can help to correct the deformity of the forefoot adduction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of recurrent idiopathic clubfoot
* The initial treatment was treated with the ponseti method
* Dynamic supination
* The max-dorsiflexion of angle <5°
* The fore foot is adduct
* The sole is cavus

Exclusion Criteria:

* Symptomatic recurrent clubfoot
* Tarsal fusion
* Rigid recurrent clubfoot

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
The adduction of foot. | Six months after the operation
  Measure the angle of foot adduction
The adduction of foot. | 1 year after operation
  Measure the angle of foot adduction

SECONDARY OUTCOMES:
The dorsiflextion of ankle. | Six months after the operation
  Measure the angle of ankle dorsiflextion
The dorsiflextion of ankle. | 1 year after operation
  Measure the angle of ankle dorsiflextion